CLINICAL TRIAL: NCT00677066
Title: A Randomised Controlled Trial: Home Oxygen Therapy Versus Hospital Oxygen Therapy for Children With Acute Bronchiolitis
Brief Title: Safety Study of Home Oxygen Therapy for Children With Acute Bronchiolitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Princess Margaret Hospital for Children (Other)
Responsible Party: Dr Andrew Martin, Princess Margaret Hospital for Children
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: EP 1405
Record Dates: First submitted 2008-05-08; First posted 2008-05-13 (Estimated); Last update posted 2008-05-13 (Estimated); Status verified 2008-05

CONDITIONS: Bronchiolitis
Keywords: bronchiolitis; oxygen; children
MeSH Terms: conditions — Bronchiolitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Children discharged home with oxygen
  Interventions: Procedure: Home oxygen therapy
- 2 (No Intervention): Children remain in hospital for oxygen therapy

INTERVENTIONS:
Procedure: Home oxygen therapy — Administer oxygen at home or in hospital
  Other Names: Home oxygen; Hospital oxygen
  Arms: 1

SUMMARY:
Home oxygen therapy is considered an appropriate and relatively safe option for children with chronic respiratory problems such as chronic lung disease of prematurity, but the use of home oxygen therapy for children with acute respiratory problems is limited. With the recent establishment of a "Hospital in The Home" (HiTH) program at our institution, we sought to determine the safety, parental satisfaction and economic advantage of home oxygen therapy for children with acute bronchiolitis compared with traditional inpatient hospitalization.

DETAILED DESCRIPTION:
Acute bronchiolitis is the most common reason for hospital admission in children aged less than 1 year in developed countries. Over the last 25 years, hospitalization rates and admission duration have increased dramatically, resulting in substantial health care costs for both institutions and individual families.

There are currently no pharmacological therapies for acute bronchiolitis that have been shown to consistently alter the natural history of this disease. Current evidence suggests that management is essentially supportive, consisting of oxygen supplementation if the child is hypoxic and nasogastric feeds or intravenous fluids if the child is dehydrated. Oxygen supplementation is the principal determinant of the length of hospital admission for children with acute bronchiolitis and the need for supplemental oxygen is generally considered to be an absolute indication for hospitalization. However, Bajaj et al demonstrated that a carefully selected population of children with acute bronchiolitis can be managed safely with home oxygen therapy.

The escalating demand and cost of health care has driven health reforms in many countries, including Australia and the United Kingdom. These reforms have included the development of services that allow patients with a range of illnesses to be managed safely in their own home rather than hospital. Such services have been well established for children with a number of chronic conditions and although managing children with acute illnesses at home is not a new strategy, this model of care is increasingly considered an alternative to traditional in-patient hospitalisation. In addition to the financial benefits of transferring care to the patients' homes for health care providers and families, children and parents report a strong preference for such models of care.

Home oxygen therapy is considered an appropriate and relatively safe option for children with chronic respiratory problems such as chronic lung disease of prematurity, but the use of home oxygen therapy for children with acute respiratory problems is limited. With the recent establishment of a "Hospital in The Home" (HiTH) program at our institution, we sought to determine the safety, parental satisfaction and economic advantage of home oxygen therapy for children with acute bronchiolitis compared with traditional inpatient hospitalization.

ELIGIBILITY:
Inclusion Criteria:

1. 3 - 24 months of age (corrected gestation)
2. Clinical diagnosis of acute bronchiolitis
3. Adequate feeding (>50% normal) & hydration
4. O2 saturation >92% on <1litre/minute nasal cannula oxygen.
5. Observed and clinically stable for at least 24 hours in hospital
6. Pass modified "safety in air test "
7. Caregivers must be counseled about risk of smoking around a child receiving oxygen supplementation
8. Caregivers must be adequately educated about home oxygen
9. HiTH nurses able to visit at home at least twice daily, in addition to daily phone call
10. Paediatrician agrees that child is eligible for recruitment in study

Exclusion Criteria:

1. Pre-existing cardiac, pulmonary (including chronic lung disease of infancy, cystic fibrosis and congenital or acquired airway anomalies), and neuromuscular disorders
2. History of apnea
3. Prematurity <34 weeks gestation

Ages: 3 Months to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 44 (Actual)
Dates: Start 2007-08; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Readmission to hospital | Within 7 days of discharge

SECONDARY OUTCOMES:
Number of days in hospital | days
parent satisfaction | discharge

CONTACTS AND LOCATIONS:
Overall Officials: Andrew C Martin, FRACP, Principal Investigator — Princess Margaret Hospital for Children
Locations (1):
- Princess Margaret Hospital for Children, Perth, Western Australia, Australia